CLINICAL TRIAL: NCT00192036
Title: Multicenter Phase II Trial Evaluating Cisplatin-Gemcitabine With Concomitant Thoracic Radiotherapy for Treatment of Inoperable Stage III Non Small Cell Lung Cancer
Brief Title: Multicenter Phase 2 Trial Evaluating Cisplatin-Gemcitabine With Concomitant Thoracic Radiotherapy for Treatment of Inoperable Stage III Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8984; B9E-BX-JHSQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-03-25 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Cisplatin (Experimental): Gemcitabine: 1250 mg/m2, intravenous (IV), day 1 and day 8 every 21 days x 3 cycles (1-3) then 300 mg/m2 x 2 cycles (4-5).
  Cisplatin: 80 mg/m2, IV, every 21 days x 5 cycles.
  Radiation: 63 Gray (Gy) in 35 treatments over 7 weeks concurrent with chemotherapy cycles 4 and 5.
  Interventions: Drug: gemcitabine; Drug: cisplatin; Radiation: radiation

INTERVENTIONS:
Drug: gemcitabine — 1250 mg/m2, intravenous (IV), day 1 and day 8 every 21 days x 3 cycles (1-3) then 300 mg/m2 x 2 cycles (4-5)
  Other Names: LY188011; Gemzar
Drug: cisplatin — 80 mg/m2, IV, every 21 days x 5 cycles
Radiation: radiation — 63 Gray (Gy) in 35 treatments over 7 weeks concurrent with chemotherapy cycles 4 and 5

SUMMARY:
The purpose of the study is to evaluate the response rate of patients with non small lung cancer to gemcitabine in combination with radiotherapy. The tolerability and safety of this combination will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable non small cell lung cancer Stage III
* Adequate hematological parameters
* Adequate Lung function reserve

Exclusion Criteria:

* Previous chemotherapy and thoracic radiation for non small cell lung cancer
* Presence of distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-08; Primary Completion 2008-01 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- Belgium (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleroi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gilly
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haine-St.- Paul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herentals
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mechelen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottignies
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turnhout

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine + Cisplatin: Gemcitabine: 1250 mg/m2, intravenous, day 1 and day 8 every 21 days x 3 cycles (1-3) then 300 mg/m2 x 2 cycles (4-5).
  Cisplatin: 80 mg/m2, intravenous, every 21 days x 5 cycles. Radiation: 63 Gray (Gy) in 35 treatments over 7 weeks concurrent with chemotherapy cycles 4 and 5.
Period: Overall Study
Arm/Group | Gemcitabine + Cisplatin
Started | 49
Completed | 28
Not Completed | 21
Not completed — Protocol Violation | 3
Not completed — Adverse Event | 6
Not completed — Patient/Physician Perception | 1
Not completed — Objective Tumor Progression | 4
Not completed — Clinical Disease Progression | 1
Not completed — Death | 1
Not completed — Unknown or Not Specified | 5

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 63.1 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 36
Region of Enrollment [Number; unit: participants]
  Belgium | 49
Basis for Pathological Diagnosis [Number; unit: participants]
  Histopathological | 39
  Cytological | 10
Disease Stage [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIA - the cancer has spread to nearby tissue or spread to near by lymph nodes. Stage IIIB - cancer spread to opposite side of chest, more than one tumor within same lobe of lung.
  participants
    Stage IIIA | 14
    Stage IIIB | 35
Karnofsky Performance Status Scale [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0-100, the lower the score, the worse the survival for most serious illnesses.
  participants
    80 - Activity with effort; some signs of disease | 9
    90 - Normal activity; minor signs of disease | 24
    100 - Normal no complaints; no evidence of disease | 16
Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma of Lung | 18
  Large Cell | 7
  Other Pathological Diagnosis | 2
  Squamous Cell | 22
Time Since Diagnosis [Mean (Standard Deviation); unit: months] | 0.5 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response at End of Treatment
Description: Response recorded at the first follow-up visit using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to first follow-up visit (up to 8 weeks after end of chemo-radiation)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49
participants
  Complete Response | 1
  Partial Response | 18
  Stable Disease | 3
  Progressive Disease | 1
  Unknown | 22
  Missing | 4

2. Secondary Outcome: Time to Progressive Disease
Description: Time to progressive disease is the time from the date of enrollment to the first date of documented disease progression. Patients who have not had disease progression will be censored at the date of the last follow-up visit. Patients dying because of reasons other than tumor progression are not included.
Time Frame: Preliminary: baseline to measured progressive disease (up to 3.5 years); Final: baseline to measured progressive disease (up to 5 years);
Population: All enrolled participants.
Measure: Median (Full Range); unit: months
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49
months
  Preliminary | 10.9 [0.9 to 39.2]
  Final | 11.4 [9.4 to 12.9]

3. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: Preliminary: baseline to date of death from any cause (up to 3.5 years); Final: baseline to date of death from any cause (up to 5 years)
Population: All enrolled participants.
Measure: Median (Full Range); unit: months
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49
months
  Preliminary | 27.9 [0.9 to 39.2]
  Final | 21.8 [17.5 to 26.0]

4. Secondary Outcome: Safety of Induction Chemotherapy
Description: A grading (severity) scale is provided for each adverse event term. Toxicities were graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) Version 2.0 grading scales. Grades range from 0 (none) to 5 (death). Number of participants with clinically significant Grade 3 and Grade 4 toxicities occurring during induction chemotherapy are reported. Grade 3 events are severe and Grade 4 events are life-threatening.
Time Frame: every cycle (21 days) for 3 cycles (up to 10 weeks)
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49
participants
  Neutropenia - Grade 3 | 9
  Neutropenia - Grade 4 | 8
  Thrombocytopenia - Grade 3 | 4
  Thrombocytopenia - Grade 4 | 1

5. Secondary Outcome: Safety of Chemo-radiotherapy
Description: A grading (severity) scale is provided for each adverse event term. Toxicities were graded according to NCI-CTC Version 2.0 grading scales. For specific radiation events, Radiation Therapy Oncology Group/European Organization for Research and Treatment of Cancer late radiation toxicity scale was used. Grades range from 0 (none) to 5 (death). Number of participants with clinically significant acute Grade 3 and Grade 4 toxicities (worst severity) occurring during chemo-radiation and up to 49 days (8 weeks) after are reported. Grade 3 events are severe and Grade 4 events are life-threatening.
Time Frame: Cycles 4 and 5 up to 8 weeks after the end of chemo-radiotherapy
Population: All enrolled participants receiving chemo-radiotherapy (Cycle 4).
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 49
participants
  Neutropenia - Grade 3 | 6
  Neutropenia - Grade 4 | 2
  Thrombocytopenia - Grade 3 | 7
  Thrombocytopenia - Grade 4 | 1
  Radiation Esophagitis - Grade 3 | 4
  Radiation Esophagitis - Grade 4 | 0
  Radiation Pneumonitis - Grade 3 | 1
  Radiation Pneumonitis - Grade 4 | 0

ADVERSE EVENTS:
Groups:
- Gemcitabine + Cisplatin: Gemcitabine: 1250 mg/m2, IV, day 1 and day 8 q 21 days x 3 cycles (1-3) then 300 mg/m2 x 2 cycles (4-5) Cisplatin: 80 mg/m2, IV, q 21 days x 5 cycles Radiation: 63 Gy in 35 treatments over 7 weeks concurrent with chemotherapy cycles 4 and 5
Arm/Group | Gemcitabine + Cisplatin
Serious Adverse Events (participants affected / at risk) | 13/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin (N=49)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hyperthermia (General disorders) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 4 (4)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Cisplatin (N=49)
Anaemia (Blood and lymphatic system disorders) | 32 (44)
Leukopenia (Blood and lymphatic system disorders) | 22 (52)
Lymphopenia (Blood and lymphatic system disorders) | 22 (34)
Neutropenia (Blood and lymphatic system disorders) | 29 (55)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (44)
Tinnitus (Ear and labyrinth disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 19 (22)
Diarrhoea (Gastrointestinal disorders) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 34 (60)
Oesophagitis (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 28 (40)
Asthenia (General disorders) | 7 (7)
Chest pain (General disorders) | 3 (3)
Fatigue (General disorders) | 21 (26)
Pyrexia (General disorders) | 5 (6)
Rhinitis (Infections and infestations) | 5 (5)
Weight decreased (Investigations) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 16 (19)
Headache (Nervous system disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 5 (6)

LIMITATIONS AND CAVEATS:
Enrollment was stopped early due to difficulties with patient recruitment. Given the number of missing/unknown tumor assessments, care should be taken when interpreting the primary outcome measure. An identified error was corrected in the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days